CLINICAL TRIAL: NCT03120455
Title: Effects of Almond Versus Pistachio on Weight Loss of Obese and Overweight Female Adults During Hypoenergetic Diet - a Randomized, 12 Week Clinical Trial
Brief Title: Effects of Almond Versus Pistachio on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-204
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Overweight
Keywords: weight loss; Almond; Pistachio; hypoenergetic diet; Nut
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Almond group (AG) (Experimental): Obese or overweight female adults will be randomly allocated to have have almond as afternoon snack while they have a hypoenergetic diet.
  Interventions: Behavioral: Almond Group
- Pistachio group (PG) (Active Comparator): Obese or overweight female adults will be randomly allocated to have have Pistachio as afternoon snack while they have a hypoenergetic diet.
  Interventions: Behavioral: Pistachio Group
- Nut Free (NFG, CG) (Placebo Comparator): Obese or overweight female adults are asked to avoid all nuts, seeds, and nut products while they have a hypoenergetic diet. , as the control group.
  Interventions: Behavioral: Nut free group

INTERVENTIONS:
Behavioral: Almond Group — Obese or overweight female adults will be randomly allocated to have almond as afternoon snacks, while they have a hypoenergetic diet.
  Other Names: AG
  Arms: Almond group (AG)
Behavioral: Pistachio Group — Obese or overweight female adults will be randomly allocated to have Pistachio as afternoon snacks, while they have a hypoenergetic diet.
  Other Names: PG
  Arms: Pistachio group (PG)
Behavioral: Nut free group — Obese or overweight female adults will be asked to avoid nuts, seeds and nut products, while they have a hypoenergetic diet.
  Other Names: NFG
  Arms: Nut Free (NFG, CG)

SUMMARY:
The purpose of the current study is comparing the effect of almond and pistachio, as the two common types of nuts, consumption on healthy obese and overweight female who following a hypocaloric diet for 12 weeks. The secondary aim of the current study is to evaluate of these two type of nuts on other cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Must be 18-45 years of age.
* Must have Body mass index (BMI) between 27-35 kg/ m².
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Have allergy to nuts
* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Weight | 12 Weeks
  Body weight was taken to the nearest 0.1 kg using a digital calibrated scale (Omron Health Care, Hoofddorp, Netherland), whilst subjects wore light clothing and no shoes.

SECONDARY OUTCOMES:
Waist circumference | 12 Weeks
  Waist circumference (WC) was measured with a rigid measuring tape and recorded to the nearest 0.5 cm. WC was measured at the smallest horizontal circumference between the ribs and iliac crest (the natural waist), or, in case of an indeterminable waist narrowing, halfway between the lower rib and the iliac crest.
fasting blood glucose | 12 Weeks
  Fasting plasma glucose (FPG) were measured using the enzymatic colorimetric method.
HbA1c | 12 Weeks
  Glycated hamoglobin (HbA1c) was measured by a colorimetric method after an initial separation by ion exchange chromatography (Biosystem, Barcelona, Spain).
HOMA-IR | 12 Weeks
  Insulin resistance was evaluated by homeostasis model assessment of insulin resistance (HOMA-IR), which was calculated by using the following formula HOMA-IR = [fasting insulin (mU/l) × FPG (mmol/l)]/22.5
lipid profiles | 12 Weeks
  Biochemical analysis of the serum total cholesterol (TC), triglyceride (TG), and high-density lipoprotein (HDL) cholesterol was carried out on a Selectra E auto analyzer (Vita Laboratory, Netherlands) following standard procedures of the Pars Azmoon diagnostic kits (Iran). The LDL cholesterol was calculated using the Friedewald formula.
  LDL cholesterol = TC - HDL cholesterol + (TG ÷ 2.2)
liver function tests | 12 Weeks
  AST ALT
Insulin | 12 Weeks
  Insulin was measured by using a radioimmunoassay with 125I-labeled human insulin and a human insulin antiserum in an immunoradiometric assay (IRMA) (Biosource, Dorest, Belgium) with a gamma-counter system (Gamma I; Genesys).

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Farshchi, MD, PhD, Study Chair — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ameneh Madjd, Dr, Principal Investigator — NovinDiet Clinic, School of Life Sciences, The University of Nottingham
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided